CLINICAL TRIAL: NCT07373119
Title: Impact of a Program Aimed at Improving Frailty in Patients With Stable Ischemic Heart Disease in Primary Care: Fragicor Study
Brief Title: Improving Frailty in Patients With Stable Ischemic Heart Disease
Acronym: FRAGICOR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ethics committee 25/198-P; Ajuts XB (Other Grant/Funding Number: Catalan Institute of Health)
Record Dates: First submitted 2025-12-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Coronary Heart Disease
Keywords: frailty; coronary heart disease; elderly
MeSH Terms: conditions — Coronary Disease; Frailty | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: It is an experimental study before-after based on a program of 12 sessions of physiotherapy in primary care setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with stable coronary heart disease (Experimental): older than 70 years, idependents in ADL
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — Primary care based physiotherapy groups

SUMMARY:
The goal of this clinical trial is to improve the frailty in old patients who have a cardiac disease .

Researchers will determine the improvement in the instability and the strength along twelve sessions based on guided exercises and mobility techniques made by physiotherapists. Research team will also evaluate the medications and diet, as well as laboratory and clinical tests.

DETAILED DESCRIPTION:
Intitial visit to measure quality of life, instability and strenght, followed by twelve sessions, one each week will be performed

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Diagnosis of coronary artery disease (International Classification Diseases (ICD)-10 I20-I25)
* Canadian Cardiovascular Society Class I
* Low cardiovascular risk according to exclusion criteria

Exclusion Criteria:

* Inability or refusal to provide informed consent (advanced dementia, severe psychiatric illness)
* Inability to perform protocol procedures
* Severe mobility-limiting conditions (Parkinson's disease, progressive neurological disorders, disabling joint disease)
* Recent (<6 months) unstable angina, myocardial infarction, coronary revascularization or angioplasty
* Deep venous thrombosis or pulmonary embolism in the last 6 months
* Recent stroke (<6 months)
* Heart failure in New York Heart Assocaition functional status (NYHA) III-IV
* Left ventricular ejection fraction < 50%
* Symptomatic valvular heart disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) components (balance, gait speed, chair rise) | From enrollment to the end of treatment ending after 12 weeks.
  Improvement in baseline values: each of the three component scores <= 4 points, and tests consists of: balance test, Gait speed and chair-stand tests. Maximum possible is 12 points and under 10 points means frailty

SECONDARY OUTCOMES:
Euroqol5D Goldberg Anxiety and Depression Scale Number of falls throughout the study Major Cardiovascular events Adherence to the program | from the baseline to 12 weeks of intervention
  Euroqol5D measures the Quality of life through an Analogic Visual Scale, which ranks from 0 (worst) to100(best) Goldberg anxiety and depression scales measure the probabilty of suffering from anxiety or depression. The tests consist in a total of 9 questions for each dimension. A score of >=4 in any of the dimensions suggest pathology.
  Adherence to the program will be evbaluated counting the attendance to the sessions. More than 9 sessions will be considerated good adherence

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Centers, Barcelona, Select..., Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form: Study protocol of Fragicor reviewed version (2026-01-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT07373119/Prot_ICF_000.pdf